CLINICAL TRIAL: NCT04969848
Title: Uncontrolled, Single-center Study to Quantify Gait Disturbance in Patients With Multiple Sclerosis
Brief Title: Quantifying Gait Alteration in Multiple Sclerosis Using a Wearable Device
Acronym: eMSGait
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0070
Record Dates: First submitted 2021-05-28; First posted 2021-07-21 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
Keywords: Wearable sensor; Gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eMSGait: Record of IGP using IMU sensor (Metamotion R mbientlab) during T25FW.
  Interventions: Other: Wearable sensor

INTERVENTIONS:
Other: Wearable sensor — IMU sensor (as part of eMSGait device) worn at the hip during T25FW
  Other Names: MetaMotionR Sensor, Mbientilab

SUMMARY:
Gait alteration is frequent in MS and limitation in walking ability is a major concern in MS patients. The development of wearable device offers the opportunity to collect data during daily activity including walking.

DETAILED DESCRIPTION:
Umanit and LMJ (Nantes university) has developed a device call eMSgait to assess walking ability in MS patients individuals (eg MS patients). This device consists in a commercialized IMU sensor (MetaMotionR Sensor, Mbientilab) worn at the right hip, a smartphone app and dedicated algorithm/mathematical model to extract raw sensor data and calculate individual gait pattern (IGP). This IGP consists of a curve, based on quaternion and representing the rotation recorded by the IMU during an average gait cycle. Pursue first pilot work assessing information from IGP on gait alteration in MS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 64 years
* Diagnosis of MS based on McDonald criteria (including Relapsing-remitting and progressive MS)
* No relapse within the last 5 weeks before recruitment
* Able to walk with or without assistance/help/aid (one or 2 canes)
* EDSS [0-6]

Exclusion Criteria:

* Women who are pregnant
* Patient having expressed their opposition
* Patient under guardianship or security measure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: MS patients cohort followed at Nantes university hospital
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Correlation with disability | One time point per patient (inclusion)
  Correlation of gait measures (mean amplitude of walking cycles (m), mean duration of walking cycles (s), Stance swing phase ratio) obtained during a walk of 25 feet with Expanded Disability Status Scale (EDSS). EDSS is an ordinal scale measuring disability and ranging from 0 (normal examination) to 10 (death due to MS) in a 0,5-point increments from score 1.

SECONDARY OUTCOMES:
Correlation with neurological function | One time point per patient (inclusion)
  Pyramidal, cerebellar and sensory functions are assessed with Kurtzke functional system scores which are based on neurological examination. Scores of the Pyramidal and sensory systems range from 0 (normal) to 6 . Cerebellar system scores range from 0 (normal) to 6. Cerebellar system scores range from 0 (normal) to 5
Correlation with gait speed | One time point per patient (inclusion)
  Timed 25-Foot Walk (T25FW). T25FW measures the time needed to complete a 25-foot walk. Two trials are averaged
Correlation with lateralization | One time point per patient (inclusion)
  Lower limb lateralization (right vs left)
Correlation with disability location | One time point per patient (inclusion)
  Upper, lower limb, trunk MS symptoms location
Correlation with MS symptoms severity | One time point per patient (inclusion)
  MS symptoms severity quote as none, mild moderate severe
Reliability of sensor measures | At the inclusion
  Gait parameters record during a 25-foot walk repeated twice at 5 min apart.
Developement of dedicated algorithm to improve signal processing from IMU. | Day 1
  Number of detected gait cycles during a foot walk.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No